CLINICAL TRIAL: NCT04362748
Title: A Phase 1 Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 256 in Patients With Advanced Solid Tumors
Brief Title: Study of AMG 256 in Adult Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20180144
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation Phase (Experimental): Determine the maximum tolerated dose (MTD) or the recommended phase 2 dose RP2D of AMG 256.
  Interventions: Drug: AMG 256
- Dose Expansion Phase: Group 1 (Experimental): Participants will be administered with the MTD or RP2D of AMG 256 identified in the dose escalation part of the study.
  Interventions: Drug: AMG 256
- Dose Expansion Phase: Group 2 (Experimental): Participants will be administered with the MTD or RP2D of AMG 256 identified in the dose escalation part of the study.
  Interventions: Drug: AMG 256

INTERVENTIONS:
Drug: AMG 256 — AMG 256 administered as an intravenous (IV) infusion.

SUMMARY:
To evaluate the safety and tolerability of AMG 256 in adult participants and to determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent prior to initiation of any study specific activities/procedures.
* Age ≥ 18 years at the time of signing informed consent.
* Life expectancy of > 3 months, in the opinion of the investigator.
* Participant must have histologically or cytologically proven metastatic or locally advanced solid tumors not amenable to curative treatment with surgery or radiation for which:
* No standard therapy exists, or
* Standard therapy has failed, not available, or
* In the investigator's opinion, standard therapy does not result in meaningful clinical benefit.
* At least 1 measurable lesion ≥ 10 mm which has not undergone biopsy within 3 months of screening scan. This lesion cannot be biopsied at any time during the study.

Exclusion Criteria:

* Primary brain tumor, untreated or symptomatic brain metastases and leptomeningeal disease.
* History of other malignancy within the past 2 years, with the following Exceptions:
* Malignancy treated with curative intent and with no known active disease present for ≥ 2 years before enrollment and felt to be at low risk for recurrence by the treating physician.
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
* Adequately treated cervical carcinoma in situ without evidence of disease.
* Adequately treated breast ductal carcinoma in situ without evidence of disease.
* Prostatic intraepithelial neoplasia without evidence of prostate cancer.
* Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ.
* History of solid organ transplantation.
* Major surgery within 28 days of study day 1.
* Live vaccine therapy within 4 weeks prior to study day 1.
* Currently receiving treatment in another investigational device or drug study, or less than 28 days since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
* Active infection requiring oral or intravenous therapy.
* Myocardial infarction within 6 months of study day 1, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or cardiac arrhythmia requiring medication.
* History of severe allergic reactions or severe acute hypersensitivity reaction.
* Female participant is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 3 months after the last dose of AMG 256.
* Female participants of childbearing potential unwilling to use 1 highly effective method of contraception during treatment and for an additional 3 months after the last dose of AMG 256.
* Female participants of childbearing potential with a positive pregnancy test assessed within 48 hours prior to day 1 of treatment by a serum pregnancy test.
* Male participants with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment and for an additional 5 months after the last dose of AMG 256.
* Male participants with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment and for an additional 5 months after the last dose of AMG 256.
* Male participants unwilling to abstain from donating sperm during treatment and for an additional 5 months after the last dose of AMG 256.
* Participant has known sensitivity to any of the products or components to be administered during dosing.
* Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the participant and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition or disease that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to participants safety or interfere with the study evaluation, procedures or completion.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | 28 days
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to 2.5 Years
Number of Participants with Treatment-Related Adverse Events | Up to 2.5 Years
Number of Participants Who Experience a Clinically Significant Change from Baseline in Vital Sign Measurement | Up to 2 Years
Number of Participants Who Experience a Clinically Significant Change from Baseline in Clinical Laboratory Tests | Up to 2 Years
Maximum Tolerated Dose (MTD) of AMG 256 | 28 days
Recommended Phase 2 Dose (RP2D) of AMG 256 | 28 days

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of AMG 256 | Up to 2.5 Years
Time to Achieve Cmax (Tmax) of AMG 256 | Up to 2.5 Years
Area Under the Plasma Concentration-time Curve (AUC) of AMG 256 | Up to 2.5 Years
Objective Response (OR) | Up to 2.5 Years
Duration of Response (DOR) | Up to 2.5 Years
Progression-Free Survival (PFS) | Up to 1 Year
Disease Control Rate (DCR) | Up to 2.5 Years
Duration of Stable Disease | Up to 2.5 Years
Overall Survival (OS) | Up to 2 Years
Number of Participants with anti-AMG 256 Antibodies | Up to 2.5 Years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (11):
- United States (4):
  - City of Hope National Medical Center, Duarte, California
  - Indiana University, Indianapolis, Indiana
  - Washington University, St Louis, Missouri
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - St Vincents Hospital Sydney, Darlinghurst, New South Wales
  - Monash Medical Centre, Clayton, Victoria
- Belgium (2):
  - Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Spain (2):
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Kroenke MA, Starcevic Manning M, Zuch de Zafra CL, Zhang X, Cook KD, Archer M, Lolkema MP, Wang J, Hoofring S, Saini G, Aeffner F, Ahern E, Cabanas EG, Govindan R, Hui M, Gupta S, Mytych DT. Translatability of findings from cynomolgus monkey to human suggests a mechanistic role for IL-21 in promoting immunogenicity to an anti-PD-1/IL-21 mutein fusion protein. Front Immunol. 2024 Jan 26;15:1345473. doi: 10.3389/fimmu.2024.1345473. eCollection 2024. PMID 38343535
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com